CLINICAL TRIAL: NCT03162016
Title: Treatment of Multiple Gingival Recession Defects Using a Xenogenic Acellular Dermal Matrix Compared to Connective Tissue Graft: a Randomized Controlled Clinical Study
Brief Title: Treatment Off Gingival Recession Defects Using a Xenogenic Acellular Dermal Matrix Compared to Connective Tissue Graft.
Acronym: MUCODERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-PP-07
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Organ Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplants of acellular matrix (Experimental)
  Interventions: Procedure: transplants
- Transplants of connective tissue (Active Comparator)
  Interventions: Procedure: transplants

INTERVENTIONS:
Procedure: transplants — Transplant of palatine tissue and transplant of connective tissue Mucoderm

SUMMARY:
Limitation of donor site and significant postoperative morbidity are often described in connective tissue graft harvesting. We want to show if mucoderm used in tunnel technique to recover miller class I and II recessions defects could be an alternative to connective tissue graft.

DETAILED DESCRIPTION:
Connective tissue graft harvested from the palate does not always have sufficient size to cover multiple recession defects. Moreover, connective tissue graft shows significant postoperative morbidity to treat generalized multiple gingival recessions. The goal of this study is to show if Mucoderm could be considered has a substitute of connective tissue graft in the coverage of gingival recession defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 45 years, postmenopausal women (ie with amenorrhea for more than a year).
* Subject with bilateral Miller class I or II recessions defects
* non smoking patients
* patients having read and understood the information note on the study and signed the informed consent form.
* patients affiliated to the social security system.

Exclusion Criteria:

* Patient with absolute contra-indication for dental surgery: valvular heart disease at risk of infectious endocarditis, recent myocardal (≤ 12 months), organ transplants, recent placement of a coronary stent (≤ 12 months), transient ischemic attacks recurrent, cardiovascular instability, uncontrolled epilepsy, rheumatic fever.
* Patient with metabolic bone disease (Paget's disease, osteomalacia, osteogenesis imperfecta)
* Patient with an ASA score ≥ 3.
* Patient with absolute contra-indication to dental surgery
* Patient with severe hematologic disease
* Patient with I or type II diabetes
* Patients with previous or current acute illness or severe chronic cardiovascular, renal, hepatic, gastrointestinal, allergic, endocrine, neuro-psychiatric, considered by the investigator to be incompatible with the conduct of the study.
* Patients treated with retinoids, oral bisphosphonates, oral anticoagulants or anticonvulsants.
* Patient have or have had cancer of the upper aerodigestive tract treated by radiotherapy.
* Patient taking a steroidal or non-steroidal anti-inflammatory, anti-cancer or immunosuppressive chemotherapy in the last 6 months.
* Patient monitoring considered difficult by the investigator.
* Patient with poor oral hygiene incompatible with oral surgery.
* Patients with periodontal disease unstabilized
* Patient with oral dermatitis or adverse occlusion.
* Patient with an acute or chronic infection of the surgical site (osteomyelitis).
* Patient with a known allergy to collagen
* Patient with autoimmune disease
* Patient with a linguistic or mental incapacity to understand information
* Patient younger than 45 years old
* Patient trust under curatorship or judicial protection
* Patients aged over 45 premenopausal.
* Patient participating in another clinical study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Root coverage | at 6 month
  Comparison of Percentage of Root coverage at baseline and 6 months postoperatively

SECONDARY OUTCOMES:
postoperation pain | at day 1 postoperation
  visual analogic scale (at control and test side),
postoperation pain | at day 2 postoperation
  visual analogic scale (at control and test side),
postoperation pain | at day 3 postoperation
  visual analogic scale (at control and test side),
postoperation pain | at day 5 postoperation
  visual analogic scale (at control and test side),
postoperation pain | at day 10 postoperation
  visual analogic scale (at control and test side),

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vincent-Bugnas S, Laurent J, Naman E, Charbit M, Borie G. Treatment of multiple gingival recessions with xenogeneic acellular dermal matrix compared to connective tissue graft: a randomized split-mouth clinical trial. J Periodontal Implant Sci. 2021 Apr;51(2):77-87. doi: 10.5051/jpis.2002400120. PMID 33913631